CLINICAL TRIAL: NCT02160275
Title: Algorithm to Control Postprandial, Post Exercise and Night Glucose Excursions in a Portable Closed Loop Format, APPEL 4
Brief Title: Algorithm to Control Postprandial, Post Exercise and Night Glucose Excursions in a Portable Closed Loop Format
Acronym: APPEL4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J.H. DeVries (Other)
Collaborators: European Commission (Other); Rijnstate Hospital (Other)
Responsible Party: Sponsor-Investigator, J.H. DeVries, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL43469.018.13
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Artificial pancreas; Bi-hormonal closed loop; Diabetes Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Loop (Active Comparator): 4 days patient-managed insulin pump therapy with blinded continuous glucose monitoring
  Interventions: Device: Insulin pump therapy
- Closed Loop (Experimental): 4 days of automated blood glucose control with the Artificial Pancreas (Inreda Diabetic BV)
  Interventions: Device: Artificial Pancreas (Inreda Diabetic BV)

INTERVENTIONS:
Device: Artificial Pancreas (Inreda Diabetic BV) — Bi-hormonal reactive closed loop system without mealtime announcement, miniaturized prototype
  Arms: Closed Loop
Device: Insulin pump therapy — Patients' own insulin pump with fast-acting insulin analog
  Other Names: Continuous subcutaneous insulin infusion
  Arms: Open Loop

SUMMARY:
In previous studies, we tested the feasibility of a bi-hormonal closed loop system. This system for automated control of blood glucose in patients with type 1 diabetes was tested in the clinical research center as well as at the home of the patients. Glucose control with automated closed loop control was comparable to patient-managed open loop control.

The closed loop system has been further developed and miniaturized (from backpack to smartphone size) in order to interfere as little as possible with daily patient life. The aim of this trial is to assess the efficacy of the new prototype at the home of the patient. It is hypothesized that the closed loop system provides better glucose control than standard open loop therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus type 1
* Treated with insulin pump therapy for a minimum of 6 months
* Age between 18 and 75 years
* Willing and able to sign informed consent

Exclusion Criteria:

* Impaired awareness of hypoglycemia (score ≥ 4) according to Gold and/or Clarke questionnaire
* BMI > 35 kg/m2
* HbA1c > 97 mmol/mol (=11.0 %)
* Use of heparin, coumarin derivatives or oral corticosteroids
* Skin condition prohibiting needle insertion
* Pregnancy and/or breastfeeding
* Living alone during the closed loop period (the patient may ask someone to stay over temporarily)
* Any condition that the local investigator feels would have interfere with trial participation or the evaluation of the results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Mean sensor glucose concentration | Day 2-4

SECONDARY OUTCOMES:
Proportion of time spent in each glycemic category | Day 2-4
  Glycemic categories:
  * Low glucose (<3.9 mmol/l and ≥ 3.3 mmol/l)
  * Very low glucose (<3.3 mmol/l and ≥ 2.8 mmol/l)
  * Dangerously low glucose (<2.8 mmol/l)
  * High glucose (> 10 mmol/l and ≤ 13.9 mmol/l)
  * Very high glucose (> 13.9 mmol/l and ≤ 22.2 mmol/)
  * Dangerously high glucose (> 22.2 mmol/l)
Number of events in each glycemic category | Day 2-4
  Glycemic categories:
  * Low glucose (<3.9 mmol/l and ≥ 3.3 mmol/l)
  * Very low glucose (<3.3 mmol/l and ≥ 2.8 mmol/l)
  * Dangerously low glucose (<2.8 mmol/l)
  * High glucose (> 10 mmol/l and ≤ 13.9 mmol/l)
  * Very high glucose (> 13.9 mmol/l and ≤ 22.2 mmol/)
  * Dangerously high glucose (> 22.2 mmol/l)
Number of carbohydrate-treated hypoglycemic events | Day 2-4
Proportion of time spent in euglycemia (≥ 3.9 mmol/l and ≤ 10 mmol/l) | Day 2-4
Glycemic variability | Day 2-4
  Calculated as Interquartile Range (IQR)
Mean sensor glucose concentration during specific periods | Day 2-4
  Periods:
  * Day
  * Night
  * Postprandial
Mean absolute relative difference between sensor values and self-monitored blood glucose values | Day 2-4
Heart rate | Day 2-4
Physical activity | Day 2-4
  Acceleration measured with a tri-axial accelerometer. The physical activity parameter is calculated as the magnitude of the total acceleration vector (square root of the sum of the squared axes).
Mean glucose concentration per day | Day 1-4
  Intervention arm (closed loop) only
Time that the control algorithm is inactive | Day 1-4
  Intervention arm (closed loop) only

OTHER OUTCOMES:
Demographic characteristics | Baseline
Weight | Baseline
Length | Baseline
Insulin use | Day 1-4
Glucagon use | Day 1-4

CONTACTS AND LOCATIONS:
Overall Officials: J. Hans DeVries, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Academic Medical Center, Amsterdam, North Holland